CLINICAL TRIAL: NCT02094755
Title: Prevalence of High On-Treatment (Aspirin and Clopidogrel) Platelet Reactivity in Patients With Critical Limb Ischemia
Brief Title: Aspirin and Clopidogrel Reactivity in Patients With Critical Limb Ischemia (CLI)
Status: Completed | Type: Observational
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Leonardo Clavijo, Assistant Professor of Clinical Medicine Director of Vascular Medicine & Peripheral Interventions, University of Southern California
Other Study IDs: D5130L00047/ISSBRIL0152
Record Dates: First submitted 2014-03-19; First posted 2014-03-24 (Estimated); Results first posted 2019-06-28 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-04

CONDITIONS: Critical Limb Ischemia
Keywords: ASA-PLAVIX Reactivity in CLI
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood Draw
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Single cohort: Single cohort will receive Blood draw only.
  Interventions: Other: Blood draw only

INTERVENTIONS:
Other: Blood draw only — Blood draw only

SUMMARY:
Critical Limb Ischemia (CLI) is defined as limb pain that occurs at rest, or impending limb loss that is caused by severe compromise of blood flow to the affected extremity. CLI is a major cause of death and disability (secondary to myocardial infarction, stroke and amputation). The mortality in patients with CLI approaches 25% and 50% at one and five years respectively. High on-treatment platelet reactivity (HPR) in patients treated with aspirin and clopidogrel (previously referred to as "resistance") is associated with an increased risk of recurrent cardiovascular events after percutaneous coronary interventions and acute coronary syndromes. The prevalence and significance of High on-treatment Platelet Reactivity (HPR) in patients with critical limb ischemia treated with aspirin and/or clopidogrel is not known.

The investigators project aims to investigate the prevalence of HPR (to aspirin and clopidogrel) in one hundred patients with diagnosis of critical limb ischemia encountered at University of Southern California (USC) affiliated hospitals (Los Angeles County Hospital and Keck Hospital of University of Southern California).

DETAILED DESCRIPTION:
This prospective clinical study will investigate the prevalence of high on- treatment platelet reactivity (HPR) in one hundred patients with critical limb ischemia (CLI), at the Keck Hospital of USC and Los Angeles County Medical Center (LAC+USC). Platelet inhibition to aspirin will be evaluated with the VerifyNow® aspirin (ASA) test. Clopidogrel platelet inhibition will be evaluated with two different tests: the vasodilator-stimulated phosphoprotein (VASP) and the VerifyNow® purigenic receptor P2Y12 (VN-P2Y12) assays. All platelet function analyses will be performed once after a minimum of one week of uninterrupted dual antiplatelet therapy with aspirin and clopidogrel. High on-treatment Platelet Reactivity on aspirin treatment (HPRA) group will be defined as aspirin reaction units (ARU) ≥550 by the VerifyNow® ASA assay. High on-treatment Platelet Reactivity on clopidogrel (HPRC) group will be defined as P2Y12 reaction units (PRU) ≥208 by the VerifyNow® assay and Vasodilator-stimulated phosphoprotein-platelet reactivity index (VASP-PRI) ≥50% by the vasodilator-stimulated phosphoprotein (VASP) assay. All other patients will be assigned to the adequate platelet reactivity on therapy (APR) group. Prevalence of high on-treatment platelet reactivity will then be calculated for aspirin and/or clopidogrel

ELIGIBILITY:
Inclusion Criteria:

* EXPERIMENTAL GROUP: Patients with a diagnosis of critical limb ischemia (CLI) and uninterrupted treatment with aspirin and/or clopidogrel for at least one week before testing.
* CONTROL GROUP: 10 normal volunteers without any known co-morbidities

Exclusion Criteria:

* Chronic use of nonsteroidal anti-inflammatory drugs, thrombocytopenia (platelet count <100 × 103/μl), use of an oral anticoagulant (warfarin), glycoprotein (GP) IIb/IIIa inhibitors, or fibrinolytic drugs within 30 days before testing. Any documented history of hypercoaguable states or history of medication non-compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The patient population will include one-hundred patients with a diagnosis of CLI. We will only include in the study CLI patients who as part of their standard of care medical treatment are receiving dual antiplatelet therapy with aspirin 81 mg and clopidogrel 75 mg daily for at least one week.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2016-11-21 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Clavijo, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Cohort
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Cohort
Number analyzed (Participants) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.2 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 50
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Asses the Prevalence of High On-treatment Platelet Reactivity in Critical Limb Ischemia Patients Treated With Aspirin and Clopidogrel.
Description: Platelet inhibition to aspirin will be evaluated with the VerifyNow® aspirin (ASA) test. Clopidogrel platelet inhibition will be evaluated with two different tests: the vasodilator-stimulated phosphoprotein (VASP) and the VerifyNow® purinergic receptor P2Y12 (VN-P2Y12) assays.
Time Frame: Single measurment after a minimum of one week of uninterrupted dual antiplatelet therapy with aspirin and clopidogrel
Population: High on-treatment platelet reactivity on clopidigrel (HPRC) was defined as VerifyNow®P2Y12 reactive units (PRU) >208 and VASP-platelet reactivity index (VASP-PRI) >50%.
  Thromboxane A2 (TXA2) inhibition was measured with the VerifyNow®aspirin test and High on-treatment reactivity on aspirin (HPRA) was defined as aspirin reaction units (ARU) >550.
Measure: Count of Participants; unit: Participants
Groups:
- Single Cohort: Patients were included who had a diagnosis of CLI and who received uninterrupted treatment with ASA and/or clopidogrel for ≥1 week prior to platelet inhibition testing.
Arm/Group | Single Cohort
Number analyzed (Participants) | 100
Participants
  HPR on Clopidogrel | 18
  HPR on Aspirin | 17
  HPR on Both | 8
  API on Both | 57

ADVERSE EVENTS:
Time Frame: Critical limb ischemia patients with clinical indication of aspirin and clopidogrel dual antiplatelet therapy with for at least 1 week as standard of care, were monitored for adverse events for the length of study participation which was 1 day from study enrollment to the last study intervention.
Description: In adherence to the clinical trials.gov adverse event and serious adverse event definitions
Arm/Group | Single Cohort
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes